CLINICAL TRIAL: NCT03348384
Title: Linking Nociceptive Opioid Peptide (NOP) Receptors With Relapse in Cocaine Use Disorders
Brief Title: [11C]NOP-1A and Cocaine Use Disorders
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Rajesh Narendran, Visiting Professor in Radiology, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO14080588; R01DA026472 (NIH)
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Cocaine Use Disorder
MeSH Terms: interventions — 3-alpha-Hydroxysteroid Dehydrogenase (B-Specific); 3-(2'-fluoro-6',7'-dihydrospiro(piperidine-4,4'-thieno(3,2-c)pyran)-1-yl)-2-(2-fluorobenzyl)-N-methylpropanamide

STUDY DESIGN:
Intervention Model Description: [C-11]NOP-1A
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cocaine use disorders (Experimental): PET scan
  Interventions: Radiation: [C-11]; Drug: NOP-1A
- Controls (Experimental): PET scan
  Interventions: Radiation: [C-11]; Drug: NOP-1A

INTERVENTIONS:
Radiation: [C-11] — Radiolabel
Drug: NOP-1A — Tracer

SUMMARY:
The goal of this study is to compared [C-11]NOP-1A binding in recently abstinent cocaine use disorders and controls.

DETAILED DESCRIPTION:
This will allow for understanding brain stress and anti-stress mechanisms that underlie abuse of cocaine in humans.

ELIGIBILITY:
[A]Cocaine use disorders

Inclusion criteria:

1. Males or Females 18-50
2. Fulfill DSM-5 Diagnosis for Cocaine use disorder
3. Medically Healthy

Major exclusion criteria:

1. Pregnancy or lactation
2. Comorbid medical, psychiatric, drug use disorders (other than cocaine, tobacco use, and recreational marijuana/alcohol use)
3. Metal implants or paramagnetic objects contained within the body which may interfere with the MRI scan
4. Currently employed as radiation worker; or participation in radioactive drug research protocols within the previous year
5. Currently on any psychotropic medications that can influence nociceptin transmission in the brain (e.g., morphine, suboxone, SSRIs, etc.)

[B] Healthy controls

Inclusion criteria:

1. Males or Females 18-50
2. Absence of present or past psychiatric conditions (including alcohol or drug use disorders)
3. A negative urine drug screen
4. Medically Healthy

Major exclusion criteria

1. Pregnancy or lactation
2. Medical, psychiatric or drug & alcohol use disorders
3. Metal implants or paramagnetic objects contained within the body which may interfere with the MRI scan
4. Currently employed as radiation worker; or participation in radioactive drug research protocols within the previous year
5. Currently on any psychotropic medications that can influence nociceptin transmission in the brain
6. Family history of a psychotic disorder, manic episode, drug use disorders in first-degree relatives.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
[C-11]NOP-1A VT | Baseline
  VT-volume of distribution expressed relative to total plasma

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No